CLINICAL TRIAL: NCT04652882
Title: A Multicenter, Double-blind, Randomized Study to Evaluate the Effects of Tasimelteon vs. Placebo in Participants With Delayed Sleep-Wake Phase Disorder (DSWPD)
Brief Title: Evaluating the Effects of Tasimelteon vs. Placebo in Delayed Sleep-Wake Phase Disorder (DSWPD)
Status: Recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Vanda Pharmaceuticals (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: VP-VEC-162-3502
Record Dates: First submitted 2020-11-19; First posted 2020-12-03 (Actual); Last update posted 2025-12-02 (Actual); Status verified 2025-11

CONDITIONS: Sleep Wake Disorders; Sleep Disorders, Circadian Rhythm; Chronobiology Disorders
MeSH Terms: conditions — Sleep Wake Disorders; Sleep Disorders, Circadian Rhythm; Chronobiology Disorders | interventions — tasimelteon

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Tasimelteon (Experimental)
  Interventions: Drug: Tasimelteon
- Placebo (Placebo Comparator)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Tasimelteon — oral capsule
  Arms: Tasimelteon
Drug: Placebo — oral capsule
  Arms: Placebo

SUMMARY:
This is a multicenter, double-blind, randomized study to evaluate the efficacy and safety of a daily single oral dose of tasimelteon and matching placebo in male and female participants with DSWPD.

ELIGIBILITY:
Inclusion Criteria:

* Ability and acceptance to provide written informed consent.
* A confirmed clinical diagnosis of Delayed Sleep-Wake Phase Disorder (DSWPD).
* Men or women between 18 - 75 years, inclusive.
* Body Mass Index (BMI) of ≥ 18 and ≤ 35 kg/m^2.

Exclusion Criteria:

* Exacerbation of an existing psychiatric condition that requires change in treatment or intervention in the past 3 months.
* Major surgery, trauma, illness, general anesthesia, or immobility for 3 or more days within the last 30 days.
* Pregnancy, recent pregnancy (within 6 weeks), or women who are breastfeeding.
* A positive test for substances of abuse.
* Current tobacco user.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 70 (Estimated)
Dates: Start 2020-12-09 (Actual); Primary Completion 2026-06 (Estimated); Study Completion 2026-06 (Estimated)

PRIMARY OUTCOMES:
Change in Sleep Onset over the treatment period, as measured by sleep diary. | 28 days

SECONDARY OUTCOMES:
Change in nighttime objective sleep-wake parameters such as sleep time, as measured by actigraphy. | 28 days
Change in nighttime subjective sleep-wake parameters such as sleep time, as measured by sleep diary. | 28 days
Assessment of safety and tolerability of daily single dose of tasimelteon, as measured by spontaneous reporting of adverse events (AEs). | 28 days

CONTACTS AND LOCATIONS:
Locations (17):
- United States (11):
  - Vanda Investigational Site, Los Angeles, California
  - Vanda Investigational Site, Redwood City, California
  - Vanda Investigational Site, Aurora, Colorado
  - Vanda Investigational Site, Boston, Massachusetts
  - Vanda Investigational Site, St Louis, Missouri
  - Vanda Investigational Site, New Hyde Park, New York
  - Vanda Investigational Site, Cincinnati, Ohio
  - Vanda Investigational Site, Cleveland, Ohio
  - Vanda Investigational Site, Columbia, South Carolina
  - Vanda Investigational Site, San Antonio, Texas
  - Vanda Investigational Site, Sherman, Texas
- Austria (2):
  - Vanda Investigational Site, Innsbruck
  - Vanda Investigational Site, Vienna
- Germany (4):
  - Vanda Investigational Site, Berlin
  - Vanda Investigational Site, Hamburg
  - Vanda Investigational Site, Marburg
  - Vanda Investigational Site, Schwerin

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Smieszek SP, Kaden AR, Johnson CE, Brzezynski JL, Xiao C, Polymeropoulos CM, Birznieks G, Emsellem HA, Polymeropoulos MH. Case report: A patient with Delayed Sleep-Wake Phase Disorder and Optic Nerve Hypoplasia treated with tasimelteon: a case study. Front Neurosci. 2023 Nov 14;17:1287514. doi: 10.3389/fnins.2023.1287514. eCollection 2023. PMID 38033548